CLINICAL TRIAL: NCT07142850
Title: A Phase I Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Intravenous Bolus and Infusion HRS-9190 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HRS-9190-102
Record Dates: First submitted 2025-08-08; First posted 2025-08-27 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-08

CONDITIONS: Skeletal Muscle Relaxation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A: Intravenous injection, 3×ED95 (Experimental)
  Interventions: Drug: HRS-9190
- Group B: Intravenous injection, 6×ED95 (Experimental)
  Interventions: Drug: HRS-9190
- Group C: 2×ED95 (intravenous bolus) + intravenous infusion (Experimental)
  Interventions: Drug: HRS-9190
- Group D: 2×ED95 (intravenous bolus) + intravenous infusion (Experimental)
  Interventions: Drug: HRS-9190

INTERVENTIONS:
Drug: HRS-9190 — HRS-9190

SUMMARY:
This study is divided into two parts. The first part adopts a single-center, randomized, single-blind, placebo-controlled dose escalation trial design to investigate the safety, tolerability, pharmacokinetics (PK), and effects on the QTc interval in healthy subjects after a single administration of HRS-9190 for injection at doses of 3 times or 6 times the ED95.

The second part uses a single-center, open-label trial design to examine the safety, tolerability, PK, pharmacodynamics (PD), and reversal effect of neostigmine (in combination with atropine) after intravenous bolus injection and continuous intravenous infusion of the loading dose (2 times the ED95) of HRS-9190 under different anesthesia regimens.

ELIGIBILITY:
Inclusion Criteria:

1. Before the trial, the subjects have been fully informed of the nature, significance, potential benefits, possible inconveniences, and potential risks and discomforts of the trial. They can understand the procedures and methods of this study, are willing to strictly abide by the requirements of the entire clinical study, and voluntarily sign the informed consent form.
2. Aged between 18 and 45 years (inclusive) at the time of signing the informed consent form, with both males and females eligible;
3. ASA physical status classification of Class I;
4. At the screening period, male subjects must weigh ≥50 kg, female subjects must weigh ≥45 kg, and the body mass index (BMI = weight (kg)/height² (m²)) is between 19 and 28 kg/m² (inclusive);
5. Female subjects of childbearing potential must agree to use highly effective contraception and avoid donating eggs from the time of signing the informed consent form until 3 months after the last dose of the investigational product. Serum pregnancy tests at the screening and baseline periods must be negative, and they must not be breastfeeding. Male subjects whose partners are females of childbearing potential must agree to use highly effective contraception and avoid donating sperm from the time of signing the informed consent form until 3 months after the last dose of the investigational product.

Exclusion Criteria:

1. Subjects with a history or current clinical acute or chronic diseases of the circulatory system, endocrine system, nervous system, digestive system, respiratory system, hematology, immunology, psychiatry, or metabolic abnormalities, who are deemed unsuitable for enrollment by the investigator;
2. Subjects with a history of neuromuscular diseases (such as myotonic dystrophy, poliomyelitis, myasthenia gravis, botulism) or a history of poliomyelitis;
3. Subjects with a history of anesthetic complications (such as a history of malignant hyperthermia or a family history of malignant hyperthermia, or those susceptible to malignant hyperthermia (patients with congenital diseases such as idiopathic scoliosis, strabismus, ptosis, umbilical hernia, inguinal hernia, etc.));
4. Subjects with a history of asthma, a history of airway diseases requiring treatment or anatomical airway abnormalities, or signs of airway abnormalities assessed during screening airway examination that may affect laryngoscope insertion or tracheal intubation;
5. During the screening or baseline period: subjects with clinically significant abnormal physical examination results as judged by the study doctor; subjects with clinically significant abnormal electrocardiograms or those with persistently/repeatedly QTcF > 450 ms in males and > 470 ms in females; subjects with hyperkalemia or hypokalemia that are judged by the investigator to be abnormal and clinically significant;
6. Subjects with a known history of allergy to the study drug or its excipients, or those with an allergic constitution (allergic to 2 or more drugs and foods);
7. Subjects who have undergone major surgery within 6 months before screening, or have a history of surgery that may significantly affect the pharmacokinetic characteristics or safety evaluation of the study drug (such as liver or kidney transplantation), or plan to undergo surgery during the trial;
8. Subjects with contraindications to the following drugs (midazolam, propofol, sufentanil, neostigmine, atropine, and sevoflurane): acute angle-closure glaucoma, allergy to eggs, egg products, soybeans or soybean products, epilepsy, angina pectoris, ventricular tachycardia, mechanical intestinal obstruction, urinary tract obstruction, arrhythmia, sinus bradycardia, hypotension, increased vagal tone, benign prostatic hyperplasia, high fever, moderate/moderate hepatic insufficiency, and the following symptoms related to halogenated anesthetics (liver dysfunction, jaundice, fever, or eosinophilia), etc.;
9. Subjects who have used any drugs that inhibit or induce hepatic drug metabolism (such as inducers-barbiturates, carbamazepine, phenytoin, glucocorticoids, omeprazole; inhibitors-SSRI antidepressants, cimetidine, diltiazem, macrolides, nitroimidazoles, sedative-hypnotics, verapamil, fluoroquinolones, antihistamines) within 1 month before drug administration;
10. Subjects who have taken antihistamines or antidepressants within 3 months before screening;
11. Subjects who have been vaccinated within 1 month before screening or plan to be vaccinated during the trial;
12. Subjects who have used any drugs or health products (including Chinese herbal medicines) within 7 half-lives or 14 days (whichever is longer) before drug administration, or who are known to may need to receive other drug treatments during the trial period as determined during screening;
13. Subjects who have participated in a clinical trial and received the trial drug within 3 months before screening, or plan to participate in other clinical trials during the trial period;
14. Subjects who have donated blood/lost ≥ 400 mL of blood (except for physiological blood loss in women), received blood transfusion or used blood products within 3 months before screening, or plan to donate blood during the trial or within 1 month after the end of the trial;
15. Subjects who smoked more than 5 cigarettes per day on average within 3 months before screening, or cannot quit smoking during the trial;
16. Subjects who drank more than 14 units of alcohol per week on average within 3 months before screening (1 unit ≈ 285 mL of beer with 3.5% alcohol content, or 25 mL of spirits with 40% alcohol content, or 85 mL of wine with 12% alcohol content), or who do not agree to abstain from alcohol during the trial;
17. Subjects who drank excessive tea, coffee, or caffeinated beverages (on average more than 8 cups per day, 1 cup = 200 mL) within 3 months before screening;
18. Subjects who consumed special foods (such as grapefruit, grapefruit juice or foods/beverages containing grapefruit juice, chocolate, tobacco, alcohol, caffeine-containing foods or beverages, etc.) within 48 hours before drug administration;
19. Subjects with positive results in one or more of the tests for hepatitis B surface antigen, hepatitis C virus antibody, syphilis, or human immunodeficiency virus antibody;
20. Subjects with a history of drug abuse or positive drug abuse screening results;
21. Subjects with positive alcohol breath screening results;
22. Subjects with difficult venous blood collection/intolerance to venipuncture, or with a history of needle phobia/blood phobia;
23. Female subjects who are pregnant or breastfeeding;
24. Subjects who may not be able to complete the study for other reasons or who are deemed unsuitable for inclusion by the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2025-08-26 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
The incidence and severity of adverse events | from ICF signing date to Day 7
Plasma histamine levels | 10 minutes before midazolam administration and 40 minutes after administration

SECONDARY OUTCOMES:
AUC0-t of HRS-9190 | 0 hour to 8 hour after administration
AUC0 inf of HRS-9190 | 0 hour to 8 hour after administration
Cmax of HRS-9190 | 0 hour to 8 hour after administration
Tmax of HRS-9190 | 0 hour to 8 hour after administration
t1/2 of HRS-9190 | 0 hour to 8 hour after administration
CL of HRS-9190 | 0 hour to 8 hour after administration
λz of HRS-9190 | 0 hour to 8 hour after administration
VZ of HRS-9190 | 0 hour to 8 hour after administration
VSS of HRS-9190 | 0 hour to 8 hour after administration
MRTinf of HRS-9190 | 0 hour to 8 hour after administration
AUC%Extrap of HRS-9190 | 0 hour to 8 hour after administration
The C-QTc relationship of HRS-9190. | At least 90 minutes before the administration of midazolam to 24 hours after the administration of the investigational product
The maximum percentage of T1 suppression | 0 hour to about 1 hour after the end of infusion
Onset time | 0 hour to about 1 hour after the end of infusion
Duration of action | 0 hour to about 1 hour after the end of infusion
Recovery time | 0 hour to about 1 hour after the end of infusion
Recovery index | 0 hour to about 1 hour after the end of infusion

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided